CLINICAL TRIAL: NCT02381847
Title: Prospective Phase III Trial Using Radical Gastrectomy With/Without HIPEC in Advanced Gastric Cancer Patients Including Adenocarcinoma of the Esophagogastric Junction
Brief Title: Radical Gastrectomy With/Without HIPEC in Advanced Gastric Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Wenxian Guan, Dean of General Surgery Department, Nanjing Drum Tower Hospital, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDTHNanjingUMS
Record Dates: First submitted 2015-02-28; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Malignant Neoplasm of Stomach
Keywords: gastric cancer; intraperitoneal chemoperfusion
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without HIPEC (No Intervention): Patients will be treated with a D2 radical gastrectomy for advanced gastric cancer and postoperative chemotherapy (SOX or XELOX).
- with HIPEC (Experimental): Patients will be treated with a D2 radical gastrectomy for advanced gastric cancer and intraperitoneal chemoperfusion with cisplatin and postoperative chemotherapy as described for the control group.
  Cisplatin: 75mg/m2 (max 150mg/m2 max 5L )
  Interventions: Procedure: intraperitoneal chemoperfusion

INTERVENTIONS:
Procedure: intraperitoneal chemoperfusion — HIPEC with cisplatin at the time of D2 radical surgery
  Other Names: HIPEC
  Arms: with HIPEC

SUMMARY:
Patients with histological proven advanced gastric cancer (including cancer of the esophagogastric junction (AEG) without evidence of distant metastases, who fulfill the inclusion and exclusion criteria, can be recruited in this study. There are two treatment groups (A and B). The D2 radical gastrectomy will be applied in both groups. Patients randomized into group B will be treated with an intraperitoneal (in the abdominal cavity) chemoperfusion with cisplatin(75mg/m2 max 150mg/m2 max 5L ). Patients randomized into group A will not accept intraperitoneal chemoperfusion. Patients in both groups receive 6 cycles of postoperative chemotherapy (SOX or XELOX) within 4-12 weeks after the surgical procedure and are followed up for 24 months.

DETAILED DESCRIPTION:
The objective of the trial is to compare the treatment of patients with advanced gastric cancer without evidence of distant metastases treated with D2 radical gastrectomy and intraperitoneal chemoperfusion (HIPEC) and postoperative chemotherapy (Group B) and patients treated with D2 radical gastrectomy alone and postoperative chemotherapy (Group A).

The hypothesis of the trial is that D2 radical gastrectomy with intraperitoneal chemoperfusion (Group B) is superior to D2 radical gastrectomy (Group A) in terms of overall survival.

The trial is designed as a prospective, randomized, open, multicenter and parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of peritoneal metastasized gastric cancer including carcinoma of the AEG.
* No evidence of distant metastases
* preoperative examination (CT/MRI) demonstrated resectable gastricc cancer with T3-T4 stage
* Written informed consent is obtained prior to commencement of trial treatment

Exclusion Criteria:

* Any previous chemotherapy or radiotherapy, and any investigational treatment for gastric cancer
* Active systemic infections
* Patients with known interstitial lung disease with New York Heart Association classification > 2
* Serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure
* cardiac arrhythmia
* Inadequate renal function at the beginning of the trial, defined as GFR less than <60 ml/min
* Inadequate liver function at the beginning of the trial, defined as Bilirubin >1.5 times ULN
* Inadequate bone marrow function at the beginning of the trial, defined as platelet count less than <150 GPT/L or neutrophil granulocyte count less than <1.5 GPT/
* Active vaccination within 6 weeks prior to randomisation
* Active hepatitis B or C infection
* Female patients who are pregnant or breast feeding
* Missing of capacity to contract
* contraindication to the drugs which are used in the trial
* Participation in another therapeutic clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | 24 months
  overall survival [ Time Frame: Death or 2 years ]

SECONDARY OUTCOMES:
complication rate | 30 days
time to progress | 24 months
  follow up every 3 months till 24 months end of study
time to distant metastasis | 24 months
  time to other distant metastases follow up every 3 months till 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wenxian Guan, Principal Investigator — China Health Ministry
Locations (1):
- Meng Wang, Nanjing, Jiangsu, China